CLINICAL TRIAL: NCT01026675
Title: Early Screening for Gestational Diabetes Mellitus
Acronym: DG2
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Principal Investigator, Jean-Luc Ardilouze, Endocrinologist, researcher, Université de Sherbrooke
Other Study IDs: 07-027; OG-3-08-2622-JA (Other Grant/Funding Number: Canadian Diabetes Association)
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women 6-13 weeks
  Interventions: Procedure: 50 g oral glucose challenge test - 75 g oral glucose tolerance test

INTERVENTIONS:
Procedure: 50 g oral glucose challenge test - 75 g oral glucose tolerance test — 50 g oral glucose challenge test at 6-13 weeks of gestation and 75 g oral glucose tolerance test at 24-28 weeks of gestation.

SUMMARY:
The working hypothesis of this proposal is that screening for gestational diabetes mellitus as early as the 1st trimester is efficient for detecting the forthcoming presence or absence of gestational diabetes mellitus. The investigators long-term goal is the prevention of gestational diabetes mellitus onset i.e. the prevention of progression to gestational diabetes mellitus, in order to enable delivery of appropriate counselling, diagnostics and treatment for pregnant women, as well as to improve pregnancy outcomes. Therefore, robust 1st trimester screening criteria is needed.

The overall objective of this proposal is to determine an accurate and valid 1st trimester 1h post 50g oral glucose challenge test plasma glucose cut-off value that is predictive of gestational diabetes mellitus onset.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yrs
* Gestational age between 6 and 13 weeks from last menstrual period,
* Alcohol < 2 drinks/day
* Not involved in regular high intensity physical activity
* Singleton pregnancy
* Otherwise good health status.

Exclusion Criteria:

* Type 1 or type 2 diabetes
* Taking drugs interfering with glucose metabolism

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant Women
Sampling Method: Non-Probability Sample
Enrollment: 1442 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
oral glucose challenge test plasma glucose value | 6-13 weeks
  the sensitivity, specificity, positive and negative predictive values of oral glucose challenge test plasma glucose >= 7.8 mmol/L during the 1st trimester (6-13 weeks of gestation), as compared with fasting 75g glucose oral glucose tolerance test performed between the 24th and 28th weeks of gestation (the Canadian Diabetes Association - CDA gold standard).

SECONDARY OUTCOMES:
oral glucose challenge test plasma glucose cut-off value | 6-13 weeks
  1st trimester 1h post 50g oral glucose challenge test plasma glucose cut-off value that offers optimal sensibility and specificity compared to the 75g oral glucose tolerance test performed between the 24th and 28th weeks of gestation, based on the ROC curve and the maximal likelihood ratio for a positive test.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Ardilouze, MD, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche clinique Étienne-Le Bel du CHUS, Sherbrooke, Quebec, Canada